CLINICAL TRIAL: NCT06090227
Title: AMPK-activation by Metformin in FSGS: AMP-FSGS
Acronym: AMP-FSGS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000035723; HT9425-23-1-0454 (Other Grant/Funding Number: Department of the Army)
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Metformin; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin + Standard of Care (Experimental): Administration of daily oral extended-release Metformin 500 mg tablets with standard of care for 6 months.
  Interventions: Drug: Metformin + Standard of Care
- Placebo + Standard of Care (Placebo Comparator): Administration of daily placebo tablets with standard of care for 6 months.
  Interventions: Other: Placebo + Standard of Care

INTERVENTIONS:
Drug: Metformin + Standard of Care — Administration of daily oral extended-release Metformin 500 mg tablets with standard of care for 6 months.
  Arms: Metformin + Standard of Care
Other: Placebo + Standard of Care — Administration of daily placebo tablets with standard of care for 6 months.
  Arms: Placebo + Standard of Care

SUMMARY:
The primary objective of this study is to determine whether extended-release MF (in addition to standard of care (S-o-C)) is superior to placebo in reducing podocyte injury and promoting podocyte survival by 6-months in Focal Segmental Glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
Focal Segmental glomerulosclerosis (FSGS) is currently the most common primary glomerular disease that progresses to ESKD in the US. FSGS is typified by significant proteinuria, and by disorganization of the actin cytoskeleton of highly specialized epithelial cells which support the glomerular capillary loop called podocytes. Podocytes are characterized by foot processes, whose disorganization with injury is visualized on electron microscopy as foot process effacement (FPE). Podocytes are also incapable of self-renewal, and podocyte loss over ~40% per glomerulus leads to proteinuria, the nephrotic syndrome (NS) and FSGS. Such critical podocyte loss alone is sufficient for progressive CKD and ESKD. Currently, the reported rate of complete and/or partial response is 40-70% in various series with a rate of progression to ESKD 30-53% in 5-10 years.

Distinct from FSGS, Minimal Change Disease (MCD), which despite showing similar diffuse FPE and NS, has preserved podocyte numbers and rare progression to ESKD (5-20% in 20 years). MCD can be morphologically indistinguishable from early FSGS, and some MCD cases reportedly transition to FSGS. Hence, identifying and targeting mechanisms in MCD that specifically promote survival of injured podocytes with FPE, could help switch an FSGS phenotype to an "MCD-like" phenotype, and prevent or retard progression of FSGS. Currently, therapeutics in FSGS focus on immune modulation, or on hemodynamic interventions used in generically all cases of NS. Specific strategies to directly promote podocyte survival and limit podocytopenia to within the critical threshold during injury, have not been pursued clinically. Hence, many FSGS cases will progress to ESKD or encounter dose limiting side-effects of immune therapies (corticosteroids, or other agents), representing a significant therapeutic gap in the field.

In this context, MF is an Ampk-activator that is widely used, demonstrably safe, and inexpensive with reported renal benefit in diabetic and non-diabetic CKD. Its specific utility to promote cell survival of injured podocytes in FSGS has never been tested. Our preclinical data shows that an "MCD-like" pathology with podocyte injury/FPE transitioned to podocytopenia and FSGS by AMPK inhibition, while AMPK activation with MF mitigated podocytopenia in FSGS models.

The purpose of this study is to test whether Metformin use in individuals with FSGS as an adjunct to standard -of-care (corticosteroids, anti RAAS measures, BP control) is safe and will activate kidney cell AMPK and reduce podocyte injury. The primary objective is to determine whether extended-release MF (in addition to standard of care (S-o-C)) is superior to placebo in reducing podocyte injury and promoting podocyte survival by 6-months in Focal Segmental Glomerulosclerosis (FSGS). Specifically, for this purpose, this study will primarily evaluate sequential urinary podocyte mRNA excretion to identify individual urinary mRNA trajectories representing podocyte injury/depletion and potential prognostic signals in the MF study limb vs control.

A secondary objective of this study is to use multiple blood, urine and biopsy assays to test whether the addition of Metformin ( to S-o-C) mitigates kidney disease progression parameters superior to placebo. These assays will include large scale urine and serum protein profiling, protein and RNA tests performed in kidney biopsies.

Another secondary objective of this study is to test whether the addition of Metformin ( to S-o-C) is safe in patients with proteinuria and FSGS. This will be accomplished by specific questionnaires and blood tests geared towards MF-associated adverse effects.

Results of this study will inform a larger, phase 2/3 randomized trial which will evaluate the efficacy of MF treatment versus placebo in attenuating proteinuria and kidney function decline in FSGS.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged greater than or equal to 18 years, but </= 80 years age at the time of signing the informed consent
4. Biopsy-confirmed primary FSGS as defined by expert renal pathology at either institutions. For homogeneity of diagnoses, demonstrable segmental or global sclerosis lesions (>/=1 glomerulus) with diffuse podocyte foot process effacement by electron microscopy (>/+ 50% of examined glomerular tufts), or show evidence of mesangial expansion or mesangial sclerosis, also confirmed by electron microscopy.
5. Therapeutic plan by treating physician for immunomodulatory treatment using Glucocorticoids.
6. Ability to take oral medication and be willing to adhere to the MF or Placebo regimen
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 12 weeks after the end of VPA administration. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner.

Exclusion Criteria:

1. Liver disease: confirmed cirrhosis liver (any stage), acute hepatitis (> 2 fold increase in liver enzymes, any coagulopathy, hyperbilirubinemia, ascites or encephalopathy)
2. estimated GFR < 32 ml/min
3. Diabetes Mellitus diagnosis at the time of biopsy or need for oral hypoglycemic agents/Insulin, or taking Metformin for other indications
4. Treatment with another investigational drug or other intervention within 3 months
5. Current pregnancy or desire to become pregnant during the study period
6. Unwilling to use two forms of birth control (for women of childbearing age)
7. Under hospice care
8. Confirmed Dementia diagnoses in EMR problem list
9. Incarceration
10. Homelessness
11. Inability to consent
12. Currently enrolled in (or completed within the past 30 days) a study of an investigational drug or device.
13. Life expectancy of less than 6 months as determined by the clinical judgement of the patient's primary physician
14. Allergy or sensitivity to Metformin
15. Platelet count < 100,000/µL; INR > 1.5; Bleeding diathesis or blood thinner use contraindicating biopsy.
16. Bleeding diathesis or blood thinner use contraindicating biopsy will be excluded entirely from participation in research biopsy portion of study only, even if anticoagulation/blood thinners can be held temporarily.
17. Simultaneous use of Carbonic anhydrase inhibitor agents
18. Use of systemic immunosuppressive medication for non-renal indications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Slope of urinary NPHS2:Creatinine ratio | 6 months following randomization
  Measure of podocinuria via evaluation of urine podocin mRNA(nphs2) (measured as number of molecules detected by qPCR in the collected urine pellet) over the creatinine concentration. Intended for evaluation of efficacy of metformin versus placebo.

SECONDARY OUTCOMES:
estimated Glomerular Filtration Rate (eGFR) | 6 months post-randomization
  Calculated from serum creatinine (mg/dl) using the CKD-EPI formula. Intended for evaluation of efficacy of metformin versus placebo.
Slope of eGFR | 6 months post-randomization
  Change in eGFR from randomization to 6 months by incorporating eGFR at all timepoints in study between baseline and 6 months post-randomization. eGFR calculated from serum creatinine (mg/dl) using the CKD-EPI formula. Intended for evaluation of efficacy of metformin versus placebo.
Urine protein:creatinine ratio | 6 months post-randomization
  Calculated ratio of urine protein and creatinine, each collected from the electronic medical record. Intended for evaluation of clinical efficacy of metformin versus placebo.
Slope of urine protein:creatinine ratio | 6 months post-randomization
  Change in urine protein:creatinine ratio from randomization to 6 months by incorporating urine protein:creatinine ratio at all timepoints in study between baseline and 6 months post-randomization. Intended for evaluation of clinical efficacy of metformin versus placebo.
Complete remission | 6 months post-randomization
  Calculated as the number of patients in complete remission, defined as <0.5 gm urine protein excretion over 24 hours, or urine protein creatinine ratio < 0.5 at 6 months post-randomization. Intended for evaluation of clinical efficacy of metformin versus placebo.
Complete or partial remission | 6 months post-randomization
  Calculated as the number of patients with complete remission (defined as <0.5 gm urine protein excretion over 24 hours, or urine protein creatinine ratio < 0.5) or partial remission (>50% reduction in proteinuria from pre-randomization). Intended for evaluation of clinical efficacy of metformin versus placebo.
Discontinuation of study drug | Within 6 months post-randomization
  Number of patients who discontinued study drug for any reason within 6 months of randomization. Intended for evaluation of patient compliance of metformin use.
Modified Kidney Disease Quality of Life (KDQOL) score | 1 month post-randomization
  Calculated as the mean (standard deviation) of all total scores. Total scores are calculated by combining scores of 8 subsections of the KDQOL, and range from 0 - 163, with higher scores representing better quality of life. Intended for evaluation of adverse effects of metformin versus placebo.
Modified Kidney Disease Quality of Life (KDQOL) score | 6 months post-randomization
  Calculated as the mean (standard deviation) of all total scores. Total scores are calculated by combining scores of 8 subsections of the KDQOL, and range from 0 - 163, with higher scores representing better quality of life. Intended for evaluation of adverse effects of metformin versus placebo.
Hypoglycemia symptom scores | 6 months post-randomization
  Calculated as the mean (standard deviation) of all total scores. Total scores are calculated by combining scores of 6 subsections of the questionnaire, and range from 0 - 18, with higher scores representing greater symptoms. Intended for evaluation of adverse effects of metformin versus placebo.
Gastrointenstinal symptom scores | 1 month post-randomization
  Calculated as the mean (standard deviation) of all total scores. Total scores are calculated by combining scores of 15 subsections of the questionnaire, and range from 0 - 105, with higher scores representing greater symptoms. Intended for evaluation of adverse effects of metformin versus placebo.
Gastrointenstinal symptom scores | 6 months post-randomization
  Calculated as the mean (standard deviation) of all total scores. Total scores are calculated by combining scores of 15 subsections of the questionnaire, and range from 0 - 105, with higher scores representing greater symptoms. Intended for evaluation of adverse effects of metformin versus placebo.
Kidney biopsy fibrosis scores | 6 months post-randomization
  Evaluation of kidney fibrosis as measured by quantification of Masson's Trichrome staining under microscopy of biopsy at 6 months post-randomization. Scores will be grouped by the following: <10%, 10-25%, 25-50%, > 50%. Intended for evaluation of clinical efficacy of metformin versus placebo.
Number of patients with Lactate levels>2.5 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Lactate levels>5 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Vitamin B12 levels <lower limit of Normal | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with serum glutamic-oxaloacetic transaminase (SGOT) >2 fold increase | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Serum Glutamic Pyruvic Transaminase (SGPT) >2 fold increase | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Serum amyloid P component (SAP) >2 fold increase | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Bililirubin-Total >2 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with Bilirubin indirect >1 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of adverse effects of metformin versus placebo.
Number of patients with hemoglobin (Hb) <9 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of disease progression and adverse effects of metformin versus placebo.
Number of patients with hematocrit (Hct) <27 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of disease progression and adverse effects of metformin versus placebo.
Number of patients with mean corpuscular volume (MCV) >100 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of disease progression and adverse effects of metformin versus placebo.
Number of patients with Total White Blood Cells (WBC) <1500 | Within 6 months post-randomization
  As determined from the electronic medical record. Intended for evaluation of disease progression and adverse effects of metformin versus placebo.
Slope of Urine Nphs2 | 6 months post-randomization
  Change in urine podocin mRNA(Nphs2), measured as number of molecules detected by qPCR in the collected urine pellet over the creatinine concentration. Slope measured by incorporating nphs2 measurements at all timepoints in study between baseline and 6 months post-randomization. Intended for evaluation of efficacy of metformin versus placebo.
Slope of Urine Aqp2 | 6 months post-randomization
  Change in urine Aquaporin-2 mRNA(Aqp2), measured as number of molecules detected by qPCR in the collected urine pellet over the creatinine concentration. Slope measured by incorporating Aqp2 measurements at all timepoints in study between baseline and 6 months post-randomization. Intended for evaluation of efficacy of metformin versus placebo.
Slope of Urine Tgfb1 | 6 months post-randomization
  Change in urine transforming growth factor-beta1 mRNA (Tgfb1), measured as number of molecules detected by qPCR in the collected urine pellet over the creatinine concentration. Slope measured by incorporating Tgfb1 measurements at all timepoints in study between baseline and 6 months post-randomization. Intended for evaluation of efficacy of metformin versus placebo.

OTHER OUTCOMES:
Body Mass Index (BMI) | 3 months post-randomization
  Measured in kg/m2. Exploratory outcome intended for evaluation of adverse effects of metformin versus placebo.
Body Mass Index (BMI) | 6 months post-randomization
  Measured in kg/m2. Exploratory outcome intended for evaluation of adverse effects of metformin versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Menon, MD, Principal Investigator — Yale University; Cijiang He, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No